CLINICAL TRIAL: NCT00708019
Title: Improving Cancer Pain Management Through Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cancer Pain Management; R01CA116423-06 (NIH)
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Cancer; Pain
Keywords: cancer pain; bone metastasis; psychoeducational intervention; nurse coaching; patient education; breast cancer
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental): Low dose of the psychoeducational intervention (i.e., 8.0 hours with the intervention nurse over 10 weeks)
  Interventions: Behavioral: PRO-SELF PLUS Pain Management Program
- High dose (Experimental): High dose of the psychoeducational intervention (i.e., 12.3 hours with the intervention nurse over 10 weeks)
  Interventions: Behavioral: PRO-SELF PLUS Pain Management Program

INTERVENTIONS:
Behavioral: PRO-SELF PLUS Pain Management Program — The psychoeducational intervention will be conducted by specially trained oncology nurses and will include the components of knowledge, skills training, and coaching to improve cancer pain management. Patients in both groups will be seen in their homes over the course of 10 weeks with phone calls conducted in between the home visits. Patients in the HIGH-DOSE group will receive 6 visits and 10 phone calls [total time 12.3 hours]. Patients in the LOW-DOSE group will receive 4 visits and 6 phone calls [8.0 hours]. Follow-up visits to assess the sustainability of the intervention will be done at 2 weeks, 1 month and 3 months after the intervention. Both quantitative and qualitative analyses will be conducted to evaluate patient outcomes.

SUMMARY:
This study will test two different doses of a psychoeducational intervention to improve cancer pain management. In addition, the study will determine if the changes in pain management behaviors that the patients and family caregivers learn continue to be used when the intervention stops. It is hypothesized that patients and family caregivers who receive the high dose intervention will have a greater decrease in pain intensity scores.

DETAILED DESCRIPTION:
Recent work from our research group demonstrated that the use of a 6-week psychoeducational intervention, called the PRO-SELF Pain Control Program, compared to standard care, resulted in clinically and statistically significant improvements in pain management in a sample of oncology outpatients with bone metastasis. While the overall effects of the intervention were significant, for approximately 70% of patients in the intervention group pain intensity scores did not decrease by > 30% and that worst pain intensity scores remained at or above 4 at the end of the intervention. Therefore, as a logical extension of this study, we propose a randomized clinical trial (RCT) that will test the effectiveness of two different doses of the revised PRO-SELF Pain Control Program [i.e., PRO-SELF PLUS-HIGH and PRO-SELF PLUS-LOW] on pain intensity and analgesic prescriptions. In addition, the sustainability of the two doses of the intervention will be evaluated. Adult oncology outpatients with pain from bone metastasis will be recruited, stratified by site and by whether or not they participate alone or with a family caregiver, and randomized to one of the doses of the intervention. The psychoeducational intervention will be conducted by specially trained oncology nurses and will include the components of knowledge, skills training, and coaching to improve cancer pain management. Patients in both groups will be seen in their homes over the course of 10 weeks with phone calls conducted in between the home visits. Patients in the HIGH-DOSE group will receive 6 visits and 10 phone calls [total time 12.3 hours]. Patients in the LOW-DOSE group will receive 4 visits and 6 phone calls [8.0 hours]. Follow-up visits to assess the sustainability of the intervention will be done at 2 weeks, 1 month and 3 months after the intervention. Both quantitative and qualitative analyses will be conducted to evaluate patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult oncology outpatients (> 18 years of age)
* able to read, write, and understand English
* agree to participate and give informed consent
* have a KPS Score of > 50
* have an average pain intensity score of > 3.0 on a 0 to 10 NRS
* have radiographic evidence of bone metastasis
* visceral or somatic pain
* have a life expectancy of at least 6 months
* are receiving outpatient treatment for cancer (not AIDS-related) with any single or combination therapy, and have a telephone line

Exclusion Criteria:

* A documented previous or current psychiatric disorder or if at the time of recruitment they are receiving hospice care in order not to interfere with the pain management program provided by hospice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Miaskowski, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - UCSF Helen Diller Comprehensive Cancer Center, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients from October 2007 to December 2012 from oncology clinics in the San Francisco Bay area.
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 92 | 93
Completed | 77 | 78
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 92 | 93 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.01 (1.19) | 59.29 (1.29) | 59.15 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 104
  Male | 39 | 42 | 81
Region of Enrollment [Number; unit: participants]
  United States | 92 | 93 | 185

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity Score
Description: Average pain was measured using a 0 (no pain) to 10 (worst pain imaginable) numeric rating scale on a daily basis.
  Change in average pain intensity between the two intervention groups was evaluated from enrollment to the end of the study (i.e., 10 weeks).
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 92 | 93
units on a scale | 1.192 [.452 to 1.932] | 1.304 [.540 to 2.069]

2. Secondary Outcome: Worst Pain Intensity Score
Description: Worst pain was measured using a 0 (no pain) to 10 (worst pain imaginable) numeric rating scale on a daily basis.
  Change in worst pain intensity between the two intervention groups was evaluated from enrollment to the end of the study (i.e., 10 weeks).
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 92 | 93
units on a scale | 1.575 [.744 to 2.375] | 1.522 [.695 to 2.349]

ADVERSE EVENTS:
Arm/Group | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/93
Other Adverse Events (participants affected / at risk) | 0/92 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No